CLINICAL TRIAL: NCT00241774
Title: Coronary Heart Disease Incidence: Depression & Inflammation Risk
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Karina Davidson, Professor of Behavioral Medicine, Columbia University
Other Study IDs: AAAA2906; R01HL080665 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In 1995, our study participants enrolled in the Nova Scotia Health Study (NSHS95). At the time of enrollment, epidemiologic data as well as blood samples were obtained. The participants have since been followed prospectively for a variety of health outcomes. We plan to assay stored blood samples collected in 1995 for markers of inflammation and link these results to existing epidemiologic and outcomes data, specifically the 7-year incidence of CAD events. Buffy coats were also obtained from the blood samples of the SAME participants for future DNA analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSHS95 samples: In 1995, our study participants enrolled in the Nova Scotia Health Study (NSHS95). At the time of enrollment, epidemiologic data as well as blood samples were obtained. The participants have since been followed prospectively for a variety of health outcomes. We plan to assay stored blood samples collected in 1995 for markers of inflammation and link these results to existing epidemiologic and outcomes data, specifically the 7- year incidence of CAD events.

SUMMARY:
To examine the associations among depression, inflammation, and coronary heart disease using an existing data base and associated plasma samples.

DETAILED DESCRIPTION:
BACKGROUND:

Classic risk factors for coronary heart disease (CHD) do not yet predict the majority of new cases. Of the novel risk factors recently explored, elevated depressive symptoms have been found in a number of prospective studies to predict new CHD cases, as have inflammatory markers, including high sensitivity C-Reactive Protein (CRP), interleukin-6 (IL-6), and intercellular adhesion molecule. Interestingly, depression and inflammatory markers have high covariation, and intervention studies indicate that reducing depression may reduce peripheral inflammation, while successfully treating inflammation may ameliorate depressive symptoms. It becomes critical then to know if these candidate CHD risk factors are independent or dependent of the other in the prediction of CHD incidence.

DESIGN NARRATIVE:

The study will determine if depressive symptoms and inflammatory markers are independent or dependent CHD risk factors, when controlling for the other known CAD risk factors. A population-based prospective study (the Nova Scotia Health Survey; NSHS95) was conducted almost 10 years ago, in which participants were randomly selected from the socialized medical registry, which includes all citizens. All classic CHD risk factors were obtained at baseline (age, sex, race, fasting lipids, diabetic status, family CHD history, resting blood pressure, exercise levels, body mass index, smoking status, and socioeconomic status). Depressive symptoms as assessed by the Center for Epidemiological Studies Depression scale were also obtained at baseline. Plasma blood samples were obtained and maintained in a -80 degree (Celsius) freezer. Participants gave permission for medical registry records to be linked to their survey data, so that objectively documented previous and future CAD events could be detected. The study will assay plasma samples for CRP, IL-6 and ICAM-1 and then statistically model the associations among depression, inflammation and CHD incidence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Able to speak English
* Enrolled in the Nova Scotia Health Study (NSHS95)

Exclusion Criteria:

* Pregnant
* Active military personnel
* Lived in Nova Scotia province for less than 3 months
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 1995, our study participants enrolled in the Nova Scotia Health Study (NSHS95). At the time of enrollment, epidemiologic data as well as blood samples were obtained. The participants have since been followed prospectively for a variety of health outcomes. We plan to assay stored blood samples collected in 1995 for markers of inflammation and link these results to existing epidemiologic and outcomes data, specifically the 7-year incidence of CAD events.
Sampling Method: Non-Probability Sample
Enrollment: 3227 (Actual)
Dates: Start 2005-08; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- See also: Primary publication — http://www.ncbi.nlm.nih.gov/pubmed/19268727